CLINICAL TRIAL: NCT02658799
Title: A Cyclic Regimen of Diclofenac Potassium May be Efficacious in the Management of Chronic Periodontitis in Adults
Brief Title: Effects of a Cyclic NSAID Regimen on Levels of GCF PGE-E2 and IL-1beta
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nilgün Özlem Alptekin, DDS, PhD, Prof, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000/071
Record Dates: First submitted 2016-01-09; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Non-steroidal Anti-inflammatory Poisoning
Keywords: periodontitis; anti-inflammatory agents
MeSH Terms: conditions — Periodontitis | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diclofenac potassium (Experimental): Cataflam (diclofenac potassium, 50 mg) b.i.d. after a meal for 6 months in a cyclic regimen.
  Administration of diclofenac potassium was undertaken from baseline to 2 months, no drug (diclofenac potassium) was administered from 2 to 4 months, then diclofenac potassium therapy was reinstituted (b.i.d.) from 4 to 6 months.
  To promote compliance, each patient was recalled monthly.
  Interventions: Drug: cataflam (diclofenac potassium)
- placebo (Active Comparator): or placebo gel caps (containing inactive filler of starch flour and carboxymethylcellulose) b.i.d. after a meal for 6 months in a cyclic regimen.
  Administration of placebo was undertaken from baseline to 2 months, no drug (placebo) was administered from 2 to 4 months, then diclofenac potassium therapy was reinstituted (b.i.d.) from 4 to 6 months.
  To promote compliance, each patient was recalled monthly.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cataflam (diclofenac potassium) — Cataflam (diclofenac potassium, 50 mg) b.i.d. after a meal for 6 months in a cyclic regimen. Administration of diclofenac potassium was undertaken from baseline to 2 months, no drug (diclofenac potassium or placebo) was administered from 2 to 4 months, then diclofenac potassium or placebo therapy was reinstituted (b.i.d.) from 4 to 6 months. To promote compliance, each patient was recalled monthly.
  Other Names: Cataflam
  Arms: diclofenac potassium
Drug: placebo — Placebo gel caps (containing inactive filler of starch flour and carboxymethylcellulose) b.i.d. after a meal for 6 months in a cyclic regimen.
  Administration of placebo was undertaken from baseline to 2 months, no drug (diclofenac potassium or placebo) was administered from 2 to 4 months, then diclofenac potassium or placebo therapy was reinstituted (b.i.d.) from 4 to 6 months. To promote compliance, each patient was recalled monthly.
  Other Names: placebo gel cap
  Arms: placebo

SUMMARY:
Non-steroidal anti-inflammatory drugs (NSAIDs) are widely used for inflammation control and pain relief. However, while adjunct use of NSAIDs is avoided for periodontal therapy because of related side effects, cyclic administration of NSAIDs may reduce or eliminate these effects. The investigators evaluated the effect of a cyclic diclofenac potassium regimen on clinical parameters and levels of prostaglandin E2 (PGE2) and interleukin-1beta (IL-1beta) in the gingival crevicular fluid (GCF) of subjects with periodontitis. Forty-one subjects with moderate to chronic periodontitis (33 men, 8 women) were divided into two groups (test and control) after initial periodontal therapy. During this 6-month, randomized, double-blind, placebo-controlled study, test (n = 28) and control (n = 13) groups were administered a cyclic regimen of diclofenac potassium (50 mg, twice daily) or placebo. Clinical measurements of disease severity and GCF sample collections were made at baseline, 2, 4 and 6 months. GCF levels of PGE2 and IL1-1beta were determined using EIA and ELISA kits, respectively.

DETAILED DESCRIPTION:
Study Design This study utilized a randomized, controlled, double-blind, parallel-group design to investigate the 6-month effect of a cyclic regimen of diclofenac potassium [50 mg, twice daily (b.i.d)] on clinical parameters of periodontal disease and levels of PGE2 and IL-1beta in GCF. After clinical and radiographic examination, subjects were divided into two groups: 28 patients in the test group and 13 patients in the control group. Of the 28 patients in the test group, ten (nine men, one woman) were smokers, eleven (six women, five men) were non-smokers, and seven (all men) were ex-smokers. Thirteen patients in the control group comprised six smokers (five men, one woman), five non-smokers (four women, one man) and two ex-smokers (both men).

Test and control groups were administered either diclofenac potassium (50 mg) or placebo gel caps (containing inactive filler of starch flour and carboxymethylcellulose), respectively, b.i.d. after a meal for 6 months in a cyclic regimen. Administration of diclofenac potassium or placebo was undertaken from baseline to 2 months, no drug (diclofenac potassium or placebo) was administered from 2 to 4 months, then diclofenac potassium or placebo therapy was reinstituted (b.i.d.) from 4 to 6 months. To promote compliance, each patient was recalled monthly. Patients in both groups were instructed on oral hygiene, including tooth brushing for at least 2 minutes (b.i.d.) and daily interdental cleaning. SRP was not carried out during these recalls. During the screening period (baseline as well as 2, 4 and 6 months), all subjects underwent physical examinations and biochemical analyses (blood chemistry, complete blood count, urinalyses and pregnancy testing).

ELIGIBILITY:
Inclusion Criteria:

* with moderate to chronic periodontal disease
* (at least two sites with loss of clinical attachment > 4mm
* alveolar bone loss of 30-50%, as judged by radiography
* received initial periodontal therapy, including scaling and root planning, as well as oral hygiene instruction less than six weeks before study commencement.

Exclusion Criteria:

* history of cardiovascular disease, renal disease, bleeding in the upper gastrointestinal tract, gastrointestinal ulcers, asthma, hypersensitivity to diclofenac or other NSAIDs, prosthetic joint replacement, or other chronic disease affecting compliance
* received antibiotics or antibacterial agents less than 6 months before study commencement
* received NSAIDs within 1 month, or phenytoin or calcium antagonists within 3 months
* history of pregnancy, lactation, or inadequate birth control

Ages: 32 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2000-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Changes in gingival crevicular fluid levels of prostaglandin E2 by 50 mg diclofenac potassium administration | Baseline, 2 months, 4 months and 6 months
  Administration of diclofenac potassium or placebo was undertaken from baseline to 2 months, no drug (diclofenac potassium or placebo) was administered from 2 to 4 months, then diclofenac potassium or placebo therapy was reinstituted (b.i.d.) from 4 to 6 months. Gingival crevicular fluid levels of prostaglandin E2 was measured by using ELISA method, at baseline, 2-month, 4-month and 6-month of the study period.
Changes in gingival crevicular fluid levels of interleukin-1beta by 50 mg diclofenac potassium administration | Baseline, 2 months, 4 months and 6 months
  administration of diclofenac potassium or placebo was undertaken from baseline to 2 months, no drug (diclofenac potassium or placebo) was administered from 2 to 4 months, then diclofenac potassium or placebo therapy was reinstituted (b.i.d.) from 4 to 6 months. Gingival crevicular fluid levels of interleukin-1beta were measured by using ELISA method, at baseline, 2-month, 4-month and 6-month of the study period.

SECONDARY OUTCOMES:
Changes in plaque index (PI) by 50 mg diclofenac potassium administration | Baseline, 2 months, 4 months and 6 months
  At baseline, 2-, 4- and 6-month, plaque index (PI) were recorded. Plaque index (PI); 0: no visible plaque, 1: minor plaque accumulation during probing, 2: visible plaque near by gingiva, 3: full plaque accumulation of the tooth.
Changes in gingival index (GI) by 50 mg diclofenac potassium administration | Baseline, 2 months, 4 months and 6 months
  At baseline, 2-, 4- and 6-month, gingival index (GI) were recorded. Gingival index (GI); 0: healthy gingiva, 1: slightly inflammation and no bleeding on probing, 2: moderate gingival inflammation and bleeding on probing, 3: spontaneous bleeding and/or suppuration.
Changes in probing depth (PD) by 50 mg diclofenac potassium administration | Baseline, 2 months, 4 months and 6 months
  At baseline, 2-, 4- and 6-month, probing depth (PD) were recorded. Probing depth (PD): with William's periodontal probe, distance between gingival margin to bottom of the sulcus).
Changes in probing clinical attachment level by 50 mg diclofenac potassium administration | Baseline, 2 months, 4 months and 6 months
  At baseline, 2-, 4- and 6-month, clinical attachment level (CAL) were recorded. Clinical attachment level (CAL); with William's periodontal probe, distance between enamel-cement junction to bottom of the sulcus).

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Füsun Oduncuoğlu, DDSPhD, Principal Investigator — Baskent University

IPD SHARING:
Plan to Share IPD: Undecided